CLINICAL TRIAL: NCT03880409
Title: How Successful is Supplemental Intraseptal Anaesthesia in Patients With Mandibular Teeth Extraction or Irreversible Pulpitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, Giath Gazal, Associate Professor, Taibah University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRB#00010037
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Overcoming the Failure of Anesthesia in the Mandibular Teeth
MeSH Terms: interventions — Lidocaine; Carticaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2% lidocaine with 1:000,000 epinephrine (Active Comparator): supplemental intraseptal injections using 0.8 mL 2% lidocaine with 1:000,000 epinephrine
  Interventions: Drug: 2% lidocaine with 1:000,000 epinephrine
- 4% articaine with 1:000,000 epinephrine (Active Comparator): buccal infiltration of 1.8 ml 4% articaine with 1:000,000 epinephrine
  Interventions: Drug: 2% lidocaine with 1:000,000 epinephrine; Drug: 4% articaine with 1:000,000 epinephrine

INTERVENTIONS:
Drug: 2% lidocaine with 1:000,000 epinephrine — 2% lidocaine with 1:000,000 epinephrine is dental local anesthesia
Drug: 4% articaine with 1:000,000 epinephrine — 4% articaine with 1:000,000 epinephrine is dental local anesthesia
  Arms: 4% articaine with 1:000,000 epinephrine

SUMMARY:
Introduction:

Local anesthetic failure is an unavoidable aspect of dental practice. A number of factors contribute to this, which may be related to either the patient or the operator. Patient-dependent factors may be anatomical, pathological or psychological1-3. Work is still going on by dental clinicians and researchers in order to find an optimal local anesthetic agent which it has a high potency and rapid onset of action.4-6. However, pain free injection also play a role in improving the patient perceptions toward the dentist and dental treatments and encouraging patients to attend a regular checkup5-8.

Failure of the local anaesthetic injections using Inferior Alveolar Nerve Block (IANB) for lower teeth in asymptomatic and symptomatic patients requires additional buck-up strategies to achieve pain free dental treatment. Otherwise, the patient complains of severe pain and hindering the clinician to proceed to the dental treatment.

Mechanism of action for intraseptal injection The route of diffusion and distribution of the anaesthetic solution in the intraseptal technique is most likely through the medullary bone (Fig. 1). It offers anaesthesia to the bone, delicate/soft tissues, root structure in the region of infusion. It is best when both pain control and haemostasis are wanted for delicate /soft tissue and bony periodontal treatment.

Figure 1: Represents the point of needle insertion for the Intraseptal Injection and the position of the needle 3mm apical to the apex of the papillary triangle5.

Advantages of intraseptal injection In contrast to IANB and local infiltration, the intraseptal technique prevents the anaesthesia of tissues such as lips and tongue hence, decreases the chances of cheek or lip biting (self-trauma). It necessitates minimum or least dosage of local anaesthetic and minimizes bleeding during the surgical procedure. This technique being less traumatic, has immediate or instantaneous (<30-sec) onset of action and comparatively less number of postsurgical complications14. Intravascular injection is extremely unlikely to occur15compared to IANB or infiltration. Assertions that intraseptal anaesthesia is immediate are properly consistent with previous clinical results. Their findings reported that the onset of action for anaesthesia was within one minute after injection. So the onset time can be considered rapid if not immediate.

Disadvantages of intraseptal Injection Clinical experience and multiple tissue punctures may be necessary to perform this technique. During the anaesthetic procedure, the anaesthetic solution may leak in to the oral cavity resulting discomfort and an unpleasant or bitter taste. The effective period anaesthesia for pulpal and soft-tissues is very limited20 hence multiple repeats may be required for longer surgical procedures.

The aim of this prospective clinical study is to determine the anesthetic efficacy of the supplemental intraseptal technique in mandibular teeth diagnosed with extraction when the conventional inferior alveolar

DETAILED DESCRIPTION:
Methods:

One hundred patients with mandibular teeth extraction will be recruited for this study. Following profound lip numbness after the administration of the conventional IAN block, dental extraction will be initiated. If patients experience moderate to severe pain during surgery either mesial and distal supplemental intraseptal injections using 0.8 mL 2% lidocaine with 1:000,000 epinephrine or buccal infiltration of 1.8 ml 4% articaine with 1:000,000 epinephrine will be administered. Success will be defined as the ability to perform surgical extraction with mild to no pain.

Patients recruited for this study will be adult patients of the College of Dentistry, The Taibah University, Almadinah Almunawwarah, who are deemed to be in good health as determined by a health history and oral questioning. All patients include in this study have to meet the following criteria: 18-65 years of age, in good health (American Society of Anesthesiologists classification I or II) and having one non-surgical tooth for extraction. Exclusion criteria were allergy to local anesthetics, history of significant medical problems (American Society of Anesthesiologists classification III or greater), having recently taken central nervous system depressants (including alcohol or any analgesic medications within 6 hours before treatment), pregnancy, lactating, or inability to give informed consent. The Taibah Dental College Human Subjects Review Committee will approve the study, and written informed consent will be obtained from each patient. After completion of the medical history and consent form, subjects completed the Modified Corah Dental Anxiety Scale Questionnaire.

To qualify for the study, patient must have a mandibular tooth (molar, premolar or anterior), which need no surgical extraction either by sectioning or raising buccal flap along with bone removal. Therefore, each patient has a tooth that fulfilled the criteria for a clinical diagnosis of non-surgical extraction. After obtaining informed consent, patients will be given IAN block and dental extraction will be initiated once the profound lower lip numbness will be felt. During the extraction process, if the patient was complaining of pain the procedure will be stopped and the patient will be asked to rate his initial pain on a 170-mm Heft-Parker visual analog scale (VAS). The VAS was divided into 4 categories as described previously. The VAS scale consists of four categories. No pain corresponded to 0 mm. Mild pain was defined as greater than 0 mm and less than or equal to 54 mm. Mild pain included the descriptors of faint, weak, and mild pain. Moderate pain was defined as greater than 54 mm and less than 114 mm. Severe pain was defined as greater than or equal to 114 mm. Severe pain included the descriptors of strong, intense, and maximum possible.

Each patient will receive a conventional IAN block using 1 cartridge of 2% lidocaine with 1:100,000 epinephrine ((Xylocaine; AstraZeneca LP, Dentsply, York, PA) using a conventional syringe (USA: ATI) and a 27-gauge, 30mm long needles (C-K Ject (27G) 0.4 x 30mm, Korea). The patient will be questioned every 2 minutes for 10 minutes or until lip numbness is apparent. Patients who do not achieve complete lip numbness within 10 minutes will disqualiﬁed from participation in the study, but dental extraction will be still performed after achieving profound anesthesia or giving additional local anesthesia.

After lip numbness, a separate buccal nerve block will be administered for the molars using a standard syringe and 0.9 mL 2% lidocaine with 1: 100,000 epinephrine.

During the extraction procedure, if the patient feel pain, the treatment will be stopped immediately, and the patient will rate his discomfort using the Heft-Parker VAS. If the pain rating is mild, extraction will continue. If the pain rating is moderate or greater (55mm or higher on the VAS), supplemental anesthesia will be administered.

The success of the IAN block will be deﬁned as the ability to carry on the tooth extraction with no or mild pain (VAS score of 0 or ≤ 54 mm, respectively). All patients experiencing moderate to severe pain upon using elevators or forceps will receive either 2% lidocaine supplemental intraseptal injections or 4% articaine buccal infiltration.

Intraseptal injections will be administered into the mesial and distal aspect of the involved tooth using 0.8 mL 2% lidocaine with 1: 100,000 epinephrine. A 27 gauge, 21mm short needle (C-K Ject (27G) 0.4 x 21mm, Korea) will be inserted into the target region which is located 2-3mm apical to the apex of the papillary triangle (Figure. 1)5. The needle is introduced into the soft tissue and advanced until contact with bone is made. Pressure must be applied to the syringe and drive the barb slightly deeper (1 to 2 mm) into the interdental septum5. Afterward, anaesthetic solution (0.4 ml) is deposited in a minimum of 20 seconds time.

Buccal infiltrations of 4% articaine (Septanest SP. Articaine hydrochloride 4% with 1:00.000 epinephrine - Septodont, France) will be administered in the muccobuccal fold of the mandibular teeth which will be extracted over 60 sec. After completion of the intraseptal injection or buccal infiltration, the dental extraction will be resumed if the patient reports no or mild pain. The patient level of pain will be assessed every 2 minutes up to 10 minutes. After 10 minutes if the patient still feels moderate to severe pain, treatment will again be stopped, and the extraction will be considered as a failure.

Injection discomfort The discomfort of the injections will be recorded by the patients following IAN block and intraseptal injections on standard 100mm visual analogue scales (VAS), tagged at the endpoints with "no pain" (0 mm) and "unbearable pain" (100 mm).

Power calculation A study with 73 patients was reported to have 84% power to detect a difference in anesthetic success rate of 30% (Webster et al, 2016) in a continuous outcome measure assuming a significance level of 5% and a correlation of 0.5 between responses from the same subject. So, a sample size of 100 patients would enable detection of a conﬁdence interval half width of 0.09 with a certainty of 90%.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age,
* In good health (American Society of Anesthesiologists classification I or II) and
* Having one non-surgical tooth for extraction.

Exclusion Criteria:

* Allergy to local anesthetics,
* History of significant medical problems (American Society of Anesthesiologists classification III or greater),
* Having recently taken central nervous system depressants (including alcohol or any analgesic medications within 6 hours before treatment),
* Pregnancy, lactating, or
* Inability to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-09 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-08 (Actual)

PRIMARY OUTCOMES:
Assessment the success of inferior alveolar nerve block during the extraction of mandible teeth will be assessed by using a 170-mm Heft-Parker visual analog scale (VAS) | 6 months
  The success of the IAN block will be deﬁned as the ability to carry on the tooth extraction with no or mild pain (VAS score of 0 or ≤ 54 mm, respectively).

SECONDARY OUTCOMES:
assessment of Injection discomfort | 6 months
  The discomfort of the injections will be recorded by the patients following IAN block and intraseptal injections on standard 100mm visual analogue scales (VAS), tagged at the endpoints with "no pain" (0 mm) and "unbearable pain" (100 mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Taibah University, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No